CLINICAL TRIAL: NCT05139290
Title: Decision-Making Experiences for Culturally Inclusive Dementia Engagement: Dyads and Families (DECIDE: Dyads and Families)
Brief Title: DECIDE: Dyads and Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kalisha Bonds Johnson, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003056; 1K23AG073516-01 (NIH)
Record Dates: First submitted 2021-11-04; First posted 2021-12-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Alzheimer Disease; Caregiver Burden
MeSH Terms: conditions — Dementia; Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: 20 dyads (PLWDs and their adult daughter caregivers) will be enrolled to participate in the behavioral intervention together.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prototype Intervention (Experimental): The prototype intervention will be likely family-based and focused on issues of communication, problem-solving, health system literacy, and family systems, all considered in the context of the African-American (AA) adult daughter role and cultural identity.
  Interventions: Behavioral: Prototype Intervention

INTERVENTIONS:
Behavioral: Prototype Intervention — The prototype intervention will be likely family-based and focused on issues of communication, problem-solving, health system literacy, and family systems, all considered in the context of the African-American (AA) adult daughter role and cultural identity.

SUMMARY:
The purpose of this study is to design and test a decision-making program that is tailored to support adult daughters making healthcare decisions for their parents who are living with memory loss to improve the quality of life of African American families.

There are two phases of this research study. The first phase will collect information by surveys and/or interviews. The surveys and interviews will ask questions about demographics (e.g., age, race/ethnicity), culture, health, family dynamics, caregiving, and healthcare experiences. The surveys will be completed by all eligible adult daughters and parents with memory loss in pairs. The interviews will be completed by a smaller number of pairs and by all former adult daughter caregivers.

The general scope of topics is caregiving experiences, cultural identity, healthcare decisions for persons living with Alzheimer's disease, and related dementias, health, and well-being. The research team will identify and examine key factors that will lead to designing and testing the feasibility of a culturally tailored prototype intervention for African American dementia dyads/families of persons living with mild to moderate Alzheimer's disease and related dementias.

DETAILED DESCRIPTION:
This is a survey/questionnaire and interview study that will examine how healthcare decisions are made for African American parents living with memory loss by African American adult daughter caregivers to develop a prototype intervention to improve how these decisions are made and improve the quality of life of African American parents living with memory loss and their African American adult daughter caregivers.

Recruitment will occur through established connections at Emory University Goizueta Alzheimer's Disease Research Center Minority Engagement Core, Emory Healthcare Integrated Memory Care Clinic, and Emory University.

Recruitment will take place in metro Atlanta and across the United States using a study flyer and video.

The flyer will include the phone number, email address of the research team, and a quick response (QR) code for potential participants to contact the research team. The video will give information about the principal investigator (PI) and the research study as a strategy to build rapport with potential participants and assuage distrust in research. Interviews will occur remotely after participants have completed the screening process and are deemed eligible for the study. This is not a no-contact study.

The data collected will be de-identified. Privacy of existing data is not a concern. This study has two phases. The first phase will consist of surveys/questionnaires and semi-structured interviews via Zoom from both the parents living with memory loss and their adult daughters as well as semi-structured interviews via Zoom of past adult daughter caregivers whose parent(s) have died or are in long-term care facilities and adult daughters caring for a parent with severe dementia only. For past adult daughter caregivers whose parents have died, the parent will need to have died at least 12 months before enrolling in the study.

In the first part of phase two (phase 2a), participants will be key informants who participate in focus group sessions using design thinking strategies to develop the prototype intervention. Key informants will consist of parent-adult daughter dyads, past adult daughter caregivers, and adult daughter caregivers of persons with severe dementia. In the last part of phase two (phase 2b), a pretest/posttest design with two follow-ups will be completed by a new set of African American parent-adult daughter dementia dyad participants. The interactions will include surveys/questionnaires and semi-structured interviews.

Data will be collected by computer/tablet and/or telephone. For participants with limited access to a computer/tablet, the surveys may be completed via paper/pencil. The general scope of topics is caregiving experiences, cultural identity, healthcare decisions for persons living with Alzheimer's disease, and related dementias, health, and well-being.

In phase one, surveys/questionnaires for persons with mild to moderate dementia will take 0.67 hours and 1 hour for adult daughter caregivers. In phase one, the semi-structured interviews will last 1 hour in total for both parent and daughter. Semi-structured interviews with past adult daughter caregivers and adult daughter caregivers of persons with severe dementia will last approximately 0.75 hours. In phase 2, key informants will have three sessions that last approximately 1.5 hours to assist with the development of the prototype intervention. In phase 2, the pretest/posttest surveys/questionnaire should last 0.33 hours for parents living with dementia and 0.67 hours for adult daughters at baseline and the 2 follow-ups. The last follow-up will consist of one semi-structured interview that will last about 0.5 hours.

Phase 1 will allow collecting and analyzing the necessary data to develop the prototype intervention that will be developed in Phase 2a and used in Phase 2b: the intervention phase.

ELIGIBILITY:
For persons living with memory loss or cognitive impairment/Alzheimer's disease and related dementias(PLWD):

Inclusion Criteria:

* self-identifies as African American
* age 50 years or older
* community-dwelling
* experiencing signs and symptoms of mild to moderate dementia through family caregiver report on the Dementia Severity Rating Scale and meeting the National Institute on Aging and the Alzheimer's Association clinical criteria for probable (Alzheimer's Disease (AD)
* able to read, speak, and understand English
* willing to participate.

Exclusion Criteria:

* any confounding significant neurologic diseases (e.g., Parkinson's) or a major psychiatric disorder (e.g., schizophrenia).

Caregiver:

Inclusion Criteria:

* self-identifies as African American
* 18 years of age or older
* daughter/daughter-in-law (including non-blood individuals)
* aids in activities of daily living and/or instrumental activities of daily living for the PLWD
* makes/takes part in formal care decisions
* able to read, speak, and understand English
* cognitively intact
* access to an internet connection
* access to a phone or computer that accepts emails.

Key informants:

Inclusion Criteria:

* Meet the criteria for PLWD and caregiver
* has experience navigating at least 2 of the following for their parent living with dementia: assisting the PLWD with getting a formal diagnosis of Alzheimer's disease and related dementias, finding/changing a healthcare provider, medication management, receiving treatment or having a procedure, conversations about hospice, palliative care, and/or end-of-life care.

Past caregiver:

Inclusion Criteria:

* Meet criteria for caregiver except not actively providing care because of the death of their parent or the parent has been transitioned to a long-term care facility.
* The death of the parent should be at least 12 months prior to recruitment.

Caregiver of persons with severe dementia

Inclusion Criteria:

- Meet criteria for caregiver except actively providing care for a parent with severe dementia based on the family caregiver report on the Dementia Severity Rating Scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Participant retention | eight weeks
  Acceptability of the intervention will be assessed with participant retention. Retention of 80% of participants from baseline to 3-month follow-up is considered successful. Attendance of dyads during program sessions during the intervention phase. The goal is to maintain ≥ 70% attendance at program sessions
Usability of Intervention | Upon completion of the intervention (estimated to be 8 weeks)
  Usability of the intervention will be assessed with a qualitative interview with the African American parent-adult daughter dyads after completing the intervention. There is not a summary score for the open-ended questions asked during the interview.
Percentage of recruitment goal achieved | Up to 6 months after the start of recruitment
  The feasibility of the intervention will be assessed as successful recruitment of study participants. This study aims to recruit 20 African American parent-adult daughter dementia dyads in ≤ 6 months. The actual recruited number of dyads will be reported as the percentage of dyads recruited within 6 months divided by 20 (actual/goal).
Change in Quality of Life-Alzheimer's Disease (QoL-AD) Scale Score | 0-month, 1 month, 3 months
  The preliminary efficacy of the intervention will be assessed with the Quality of Life-Alzheimer's Disease (QoL-AD) scale. The QoL-AD has 13 items which are scored as poor = 1, fair = 2, good = 3, excellent = 4. The total score ranges from 13 to 52 and higher scores indicate a greater quality of life.
Change in Decision Self-Efficacy Scale Score | 0-month, 1 month, 3 months
  The preliminary efficacy of the intervention will be assessed with the Decision Self-Efficacy Scale. The Decision Self-Efficacy Scale has 11 items which are scored as not at all confident = 0 to very confident = 5. The total score ranges from 0 to 100 and higher scores indicate greater self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Kalisha Bonds Johnson, PhD RN PMHNP, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Zeta Phi Beta Sorority, Inc., Washington D.C., District of Columbia
  - Emory Healthcare Integrated Memory Care Clinic, Atlanta, Georgia
  - Emory University Goizueta Alzheimer's Disease Research Center Minority Engagement Core, Atlanta, Georgia
  - Metro-Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Researchers will share demographic data, study measures, and outcome variables
Supporting Information: Study Protocol
Time Frame: six months after publication.
Access Criteria: Researchers will share the data with qualified researchers who complete a formal data sharing agreement for research purposes only.

REFERENCES:
- [Derived] Bonds Johnson K, Lyons KS, Epps F, Daniel G, Monin JK, Powell W, Hepburn K. Development and evaluation of a healthcare decision-making intervention for African American parent-adult daughter dementia dyads: a mixed-methods study protocol. BMJ Open. 2025 Mar 13;15(3):e099976. doi: 10.1136/bmjopen-2025-099976. PMID 40081986